CLINICAL TRIAL: NCT06285253
Title: A Phase 1 Prospective Study of the Miromatrix External Liver Assist Product (miroliverELAP®) for Liver Support in Adults With Acute Liver Failure.
Brief Title: miroliverELAP® for the Treatment of Acute Liver Failure: A Phase 1 Trial
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Miromatrix Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRO-01-001
Record Dates: First submitted 2024-02-21; First posted 2024-02-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Acute Liver Failure; Acute Liver Injury, Drug Induced; Acute on Chronic Liver Failure (ACLF); Acute Alcoholic Hepatitis
Keywords: Acute liver failure; Extracorporeal liver assist; Bioengineered liver
MeSH Terms: conditions — Liver Failure, Acute; Chemical and Drug Induced Liver Injury; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Intervention Model Description: Single arm, open label, safety study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- miroliverELAP treatment (Experimental): 48 hour treatment with miroliverELAP
  Interventions: Combination Product: miroliverELAP treatment

INTERVENTIONS:
Combination Product: miroliverELAP treatment — Subject's blood will be perfused through a bioengineered liver graft via an extracorporeal blood circuit.

SUMMARY:
The clinical trial will assess the safety of miroliverELAP for the treatment of acute liver failure, severe acute alcohol-associated hepatitis, or acute on chronic liver failure. miroliverELAP is an external liver assist combination product consisting of a single-use MIRO-001 bioengineered liver graft and an extracorporeal blood circuit. miroliverELAP Is intended to support the native (failed) liver for up to 48-hours of continuous treatment to allow time for liver recovery or to identify a transplantable liver.

DETAILED DESCRIPTION:
This is a phase 1, open, single arm safety study of miroliverELAP for the treatment of acute liver failure (ALF), severe acute alcohol-associated hepatitis, or acute on chronic liver failure . Subjects who present with ALF, severe acute alcohol-associated hepatitis, or acute on chronic liver failure may be eligible for the study. Subjects will be treated with miroliverELAP continuously for 48 hours. The study will assess the safety of the miroliverELAP used to support liver function in an individual experiencing ALF, severe acute alcohol-associated hepatitis, or acute on chronic liver failure. Safety profile will be characterized by survival over the duration of therapy, tracking miroliverELAP-related adverse events, the proportion of subjects surviving 21-day post treatment initiation, and the difference in the values of specific biomarkers pre-treatment and at the time of treatment discontinuation; such as: albumin, ammonia, creatinine, INR, and lactate blood concentration. A minimum of 5 subjects will be treated for 48 hours and followed for 32 days. Up to 15 subjects may be enrolled in up to 8 study sites.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years to 80 years old at the time of signing the informed consent
2. Subject must:

   1. be deemed competent to consent by an independent qualified practitioner, or
   2. have consent given by a Legally Authorized Representative
3. Subject should be in the intensive care unit
4. Be diagnosed with 4.1. Acute Liver Failure defined as:

   1. INR ≥ 2.0, and
   2. Hepatic Encephalopathy Grade II-III (West Haven Criteria), and
   3. Less than 4 weeks (28 days) of disease duration 4.2. Severe Acute Alcohol-Associated Hepatitis as defined as:

   <!-- -->

   1. Hepatic Encephalopathy Grade I-III (West Haven Criteria), and
   2. Model for End-Stage Liver Disease (MELD) Score ≥ 20, and
   3. INR ≥ 2.0, and
   4. No overt evidence of cirrhosis 4.3. Acute on Chronic Liver Failure:

   <!-- -->

   1. Hepatic Encephalopathy Grade I-III (West Haven Criteria), and
   2. Model for End-Stage Liver Disease (MELD) Score ≥ 20, and
   3. INR ≥ 2.0,

      5. Subject is not a candidate for liver transplant and will not become a candidate in the event of worsening conditions.

Exclusion Criteria

1. Grade IV West Haven Encephalopathy Criteria
2. Previous liver transplant
3. Currently requires chronic hemodialysis (CRRT or other forms of continuous renal replacement are allowed).
4. Uncontrolled documented infection, hypotension, or refractory shock. This is defined as a need for a single vasopressor, or combination of vasopressors, that exceed a norepinephrine equivalent of 0.5 mcg/kg/min.
5. Liver injury due to trauma
6. Any current liver cancer
7. Currently on medications with a narrow therapeutic index
8. Platelet count < 40,000 μL
9. If the subject is intubated and has an acute lung injury
10. Experiencing a bleeding event, defined as:

    1. Active gastrointestinal or other overt bleeding event, or
    2. Hemoglobin drop > 3g/dL within the past 24 hours, or
    3. Received ≥ 3 units of red blood cell transfusion within the past 24 hours
11. Female that is currently pregnant, planning to be pregnant, or currently breastfeeding
12. Refusal to receive blood products

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 48 hours
  Survival over the duration of miroliverELAP treatment
Adverse Events | 32 days
  Serious adverse events attributable to miroliverELAP

SECONDARY OUTCOMES:
21-day survival | 21 days
  Survival for 21-days post initiation of miroliverELAP therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jack Lake, MD, Study Chair — Miromatrix
Locations (8):
- United States (8):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Michigan Medical School, Ann Arbor, Michigan
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Recanati/Miller Transplantation Institute, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Intermountain Healthcare, Salt Lake City, Utah
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No